CLINICAL TRIAL: NCT06059469
Title: PRISMA: A Single-centre, Prospective Phase II Imaging Study Using PSMA-PET/CT to Assess the Expression of Specific Membrane Antigen (PSMA) in Patients With Progressive Triple-negative Breast Cancer.
Brief Title: PSMA-PET/CT to Assess the Expression of Specific Membrane Antigen (PSMA) in Patients With Progressive Triple-negative Breast Cancer.
Acronym: PRISMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJBMNdTNBC
Record Dates: First submitted 2023-09-06; First posted 2023-09-28 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with progressive metastatic TNBC and presenting measurable disease on 18F-FDG PET/CT (Experimental): Patients with progressive metastatic TNBC and presenting measurable disease on 18F-FDG PET/CT
  Interventions: Diagnostic Test: Ga-PSMA PET/CT

INTERVENTIONS:
Diagnostic Test: Ga-PSMA PET/CT — Patient undergo Ga-PSMA PET/CT prior to the start of the new drug treatment

SUMMARY:
This is a descriptive, prospective, single centre study. This study will assess PSMA expression via the uptake of radiolabelled PSMA-ligand using PET/CT imaging in mTNBC lesions pre-identified on 18F-FDG PET/CT in order to evaluate the feasibility of molecular radionuclide therapy in refractory mTNBC using the Lutetium-177 radiolabelled PSMA.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with institutional guidelines and obtained prior to any study procedure
* Women with ≥ 18 years-old
* Eastern Cooperative Oncology Group Performance Status of 0 to 2
* Confirmed diagnosis of progressive metastatic TNBC and presenting measurable disease on 18F-FDG PET/CT (performed within 2 weeks) or Brain MRI in case of progressive brain metastases (performed within 4 weeks) prior to PSMA PET/CT.
* Radiolabelled PSMA PET/CT has to be performed before the next treatment line initiation

Exclusion Criteria:

* Pregnant or lactating patients
* Other active neoplastic disease
* Treatment by another molecule that is the object of investigation within 30 days
* Skin only metastatic disease
* Patients with a significant medical, neuro-psychiatric, or surgical condition, which, in the investigator's opinion, may interfere with completion of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with ≥ 18 years-old
Enrollment: 20 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess PSMA expression in progressive metastatic TNBC patients | once at baseline prior to the start of the new anti cancer treatment
  uptake of radiolabelled PSMA-ligand in patients with mTNBC on PET/CT images.

SECONDARY OUTCOMES:
Assess the concordance between lesions visualized on PSMA PET/CT and 18F-FDG PET/CT images (or brain MRI in case of brain metastases). | once at baseline prior to the start of the new anti cancer treatment
  Matching between FDG and PSMA-labelled radiotracers uptake: on PSMA PET/CT and 18F-FDG PET/CT images, each lesion will be identified and faced with the other images. Each imaging pair will be classified as complete match, partial match or no match between the different types of imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium